CLINICAL TRIAL: NCT05028842
Title: Effect of Lockdown During COVID 19 Pandemic on Liver Disease and Metabolic Parameters.
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-COVID-06
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non Cirrhotic: Non Cirrhotic
  Interventions: Other: No intervention
- Compensated Cirrhotics: Compensated Cirrhotics
  Interventions: Other: No intervention
- Decompensated Cirrhotics: Decompensated Cirrhotics
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — None.This is an observational study

SUMMARY:
The novel corona virus disease (COVID-19), pandemic has costed lives of several hundred thousands and affected millions. Comorbidities such as metabolic syndrome components and chronic liver disease have been associated with more severe infection and increased risk of death in this pandemic. Several measures have been taking by the governments across the world. An important step taken by the Indian government was the temporary lockdown of the whole country starting from 25th March 2020 till 31st May. This was followed by relaxation in phases across the country. Lockdown and social distancing helped in controlling the pandemic, but had enormous impact on health of non-COVID patients, economics and social life. Impact of lockdown COVID-19 on metabolic control in type 2 diabetes mellitus and healthy people is studied. However, the impact on liver disease patients is not known.

DETAILED DESCRIPTION:
Aim and Objective -

* Primary objective: Change in liver stiffness measured by fibroscan before and after implementation of lockdown in patients of liver disease without COVID-19 infection.
* Secondary objectives: Change in liver fat content measured by fibroscan as Controlled Attenuation Parameter (CAP) value, metabolic and laboratory parameters.

  (b) Methodology: OPD records of all consecutive patients of liver disease without COVID-19 infection from the Institute database from 1st January 2020 attending the liver clinic till 31st December 2020 will be reviewed. Patients with atleast two OPD visits, with one before implementation of lockdown and the other during the lockdown phase will be analysed. Patients of liver disease without atleast 2 fibroscan examination (one before lockdown and the other after lockdown implementation) will be excluded. In patients having more than one lockdown OPD visit, the one done at later time will be taken into consideration.
* Study population: Patients of liver disease attending the OPD with one visit before implementation of lockdown and the other during the lockdown phase.
* Study design: Retrospective
* Study period: NA
* Monitoring and assessment: OPD records of patients fulfilling the inclusion / exclusion criteria will be analysed for liver stiffness and CAP using Fibroscan, body weight, body mass index (BMI), complete blood count (CBC), liver function tests (LFT), kidney function test (KFT), HbA1c, fasting blood glucose, post prandial blood glucose, total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides.
* Statistical Analysis: Baseline parametric data will be expressed as the proportion, mean± standard deviation and median with interquartile range. Categorical variables will be analyzed by chi squared test or Fisher exact test while the continuous variables will be analyzed using unpaired t-test or Mann-Whitney test as appropriate. Paired t-test will be used to compare the change before and after the intervention. The p value < 0.05 will be considered statistically significant.
* Adverse effects: NA
* Stopping rule of study: NA

Expected outcome of the project: Results of the study will be helpful in analyzing its impact on liver and metabolic health in liver disease patients. Importance of adequate compliance to the pharmacotherapy and healthy life style will be highlighted if result shows negative impact as the pandemic is still far from over.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of liver disease attending the OPD.

Exclusion Criteria:

1. Patients without atleast 2 fibroscan examination (one before lockdown and the other after lockdown implementation).
2. Acute self-limiting hepatitis.
3. Sick patients requiring hospital admission.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of liver disease attending the OPD with one visit before implementation of lockdown and the other during the lockdown phase
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Change in liver stiffness measured by fibroscan before and after implementation of lockdown in patients of liver disease without COVID-19 infection | Day 0

SECONDARY OUTCOMES:
Change in liver fat content measured by fibroscan as Controlled Attenuation Parameter (CAP) value | Day 0
Change in weight | Day 0
Change in BMI | Day 0
Change in Liver Function tests | Day 0
Change in CBC | Day 0
Change in Fasting Blood Sugar | Day 0
Change in HbA1c | Day 0
Change in Lipid Profile | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided